CLINICAL TRIAL: NCT03412461
Title: Bridging the Gap - Tools for Finding Health, Mental Health and Wellness Resources for University and College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, David Wiljer, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 023/2017
Record Dates: First submitted 2017-11-03; First posted 2018-01-26 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Adolescent; Mental Health Wellness 1; Self Efficacy; Stigma, Social
Keywords: Transition-aged youth; Mental Health; Accessibility
MeSH Terms: conditions — Social Stigma; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Students will be recruited and randomized to the intervention arm or the control arm. The intervention group participants will have access to the Thought Spot platform. The control group participants will receive a pamphlet that outlines mental health services and wellness services across the GTA. Both groups will also have access to usual care.
Who Masked: Participant, Investigator
Masking Description: To maintain partial blindness, researchers administering surveys will not be aware of the group allocation of participants. A researcher who will not be in contact with participants will conduct the randomization. Recruitment materials do not include any reference to the intervention (Thought Spot) and therefore, mitigates any potential demand characteristics among participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thought Spot Application (Experimental): Participants randomly assigned to the experimental arm will have access to the Thought Spot application. The Thought Spot application is a mobile app and website. This digital platform was designed and produced in partnership with transition aged youth in post-secondary education. The platform maps out wellness and mental health services across the Greater Toronto Area. This group will continue to have access to usual care.
  Interventions: Other: Thought Spot
- Resource pamphlet (Active Comparator): Participants randomly assigned to the active comparator will receive a pamphlet that outlines mental health services and wellness services across the Greater Toronto Area. This group will continue to have access to usual care.
  Interventions: Other: Resource Pamphlet

INTERVENTIONS:
Other: Thought Spot — Thought Spot is a mobile app and website. This digital platform was designed and produced in partnership with transition aged youth in post-secondary education. The platform maps out wellness and mental health services across the Greater Toronto Area.
  Arms: Thought Spot Application
Other: Resource Pamphlet — The resource pamphlet that participants will be given will include information on the mental health and wellness services available at their respective post-secondary institution.
  Arms: Resource pamphlet

SUMMARY:
Background: Seventy percent of lifetime cases of mental illness emerge prior to age 24. While early detection and intervention can address approximately 70% of child and youth cases of mental health concerns, the majority of youth with mental health concerns do not receive the services they need.

Objective: This project will evaluate the impact of Thought Spot upon intentions and self-efficacy in help-seeking for mental health concerns among transition aged youth (youth aged 17-29) enrolled full-time or part-time at a college or university in the Greater Toronto Area (GTA), compared with a control group (who receive usual care; resource pamphlet).

Methods: A two-group partially blinded pre-post randomized controlled study will be done to evaluate the impact of the digital platform, Thought Spot, on transition-aged youths' intentions to help-seek. Measurements will be taken over a 6 month period: baseline, 3 months, and 6 months. 472 participants who are enrolled part-time or full-time at one of 3 participating post-secondary institutions (George Brown College, Ryerson University, University of Toronto) who are interested in maintaining or managing their mental health will be recruited and randomized to the intervention arm or the control arm. The intervention group participants will have access to the Thought Spot platform. The control group participants will receive a pamphlet that outlines mental health services and wellness services across the GTA. Both groups will also have access to usual care.

Results: The investigators are testing the hypothesis that 1) transition-aged youth who receive the intervention will show a greater improvement in intentions and self-efficacy in help-seeking for mental health concerns than those who are allocated to the control group; and 2) participants in the intervention arm will also show greater improvements in health literacy, including awareness of available services and supports, increased self-efficacy in managing their mental health concerns, and a reduction in mental health stigma, compared to the control arm.

DETAILED DESCRIPTION:
This study is an innovative randomized control trial, in its testing of a youth-driven mHealth (mobile health) intervention for its effectiveness. The study will extend and advance our understanding of whether mHealth (mobile health) interventions can help bridge the health literacy gap, facilitate increased self-efficacy and lead to enhanced help-seeking abilities for the target population. This study is a two-group partially blinded pre-post randomized controlled study to evaluate the impact of the digital platform, Thought Spot, on transition-aged youths' self-efficacy in help-seeking. Measurements will be taken over a 6 month period: baseline, 3 months, and 6 months. 472 participants who are enrolled part-time or full-time at one of 3 participating post-secondary institutions (George Brown College, Ryerson University, University of Toronto) who are interested in maintaining or managing their mental health will be recruited and randomized to the intervention arm or the control arm. 236 subjects will be recruited for the intervention arm and 236 subjects for the control arm at baseline. The intervention group participants will have access to the Thought Spot platform (study tool #1). The control group participants will receive a pamphlet that outlines mental health services and wellness services across the GTA (Greater Toronto Area) (study tool #2). Both groups will also have access to usual care including access to campus health services for mental health and wellness and web- and print- based information materials. Data will be collected from participants through a battery of online questionnaires to measure primary outcomes (changes in help-seeking intentions), help-seeking behaviours and help-seeking attitudes (secondary outcomes) as well as self-reported changes in self-stigma and self-efficacy, data on demographics and general mental health status. A final usabilitiy survey will be administered to participants in the intervention arm at the 6-month mark, followed by a purposeful sample of 15-20 of these participants for qualitative interviews to further explore usability related to app acceptance, feasibility and performance. This extra step will be done after the last survey package has been administered and should not influence or confound results since both study arms will be receiving the exact same treatment and completing the exact same sets of surveys up to this point. Digital data from the Thought Spot platform will be used to expand on the self-report data collected from participants through the various scales and measures. Participants will receive a small compensation for completion of the study (completing all three surveys) to minimize overall attrition.

Objectives Primary objective: To evaluate the impact of Thought Spot upon intentions in help-seeking for mental health concerns among transition aged youth (youth aged 16-29) enrolled full-time or part-time at a college or university in the GTA, compared with a control group (who receive usual care; resource pamphlet).

Secondary objective: To examine whether participants in the intervention arm will show greater improvements in health literacy, including awareness of available services and supports, increased self-efficacy in managing their mental health concerns, and a reduction in mental health stigma, compared to the control arm.

Data Analysis Statistical Analyses All analyses will be carried out using SAS System 9.4 for Windows. Statistical tests will be 2 sided, with confidence levels of 0.05. Prior to testing, a series of univariate analyses will be carried out to ensure that model assumptions are met. To address the primary study hypothesis, a mixed-effect model will be used to account for the longitudinal nature of the data, and for attrition. Missing values will be treated with maximum likelihood estimation in SAS PROC MIXED, which uses all available information in the data. Intention-to-treat analysis will be used; all patients will be analyzed as they were originally allocated after randomization. As a sensitivity analysis, the final model will be fitted only with subjects for whom there is complete data. Formal help-seeking score will be the dependent variable, with study groups (intervention and control) and time points as predictors, and relevant socio-demographics collected at baseline as covariates to control for possible confounding.

The interaction between study group and time will be included in the model, and linear contrasts will be used to compare the groups, specifically regarding the change from baseline to the final time point. Similar models will be used to address the exploratory hypotheses, which examine different scales and trends, on the effect of the intervention over time. Bonferroni adjustment will be used to control the Type I error rate if multiple comparisons are desired. Generalized estimating equations will be used for the Actual Help Seeking Questionnaire (AHSQ), since this scale is binary.

Other Analyses A sex- and gender-based analysis will be completed when analyzing data for Phases 1 and 2. An economic evaluation of the Thought Spot intervention compared to usual care will also be explored to determine the potential cost-effectiveness and financial implications of sustainable and widespread use of Thought Spot throughout Canadian postsecondary campuses. The evaluation will be conducted from the perspective of future potential Thought Spot funders (eg, other Canadian postsecondary institutions). The primary outcome to be assessed will be the change in helping-seeking intentions among the target population

A cost-effectiveness analysis will be conducted to compare the cost and outcome of the intervention arm against usual care. The main output will be an incremental net benefit of the intervention compared to usual care [39] and an incremental cost for one point improvement in the General Help Seeking Questionnaire (GHSQ) in a form of an incremental cost-effectiveness ratio. The investigators will characterize the uncertainty of the findings using 95% confidence interval and a cost-effectiveness acceptability curve.

Digital data collected from the Thought Spot app will be collected and analyzed to expand on the self-report data collected from participants through the various scales and measures. Usage metrics outlining the intensity of use, usage of content, and methods of accessing app data will be calculated and analyzed. Simple descriptive statistics will also be used to report the time spent on specific app features; number of times the app is used in a day; what times in the day features are being used; and number of added spots, thoughts, and reviews. We will also conduct a high-level text analysis of the added reviews of services. This has the potential to inform a scoping review on what transition aged youth what from services. Data collected from reviews can provide the researchers with a clearer idea of what students and youth want from mental health and wellness services.

Usefulness, satisfaction, ease of use, acceptance, feasibility and performance will be analyzed through the end-of-study usability survey. Results will be analyzed using means and standard deviations of all respondents for each category of the questionnaire. The proportions of participants reporting high, medium, or low levels of satisfaction will also be calculated. The open-ended survey questions will be analyzed thematically. The findings may be correlated with the other study surveys and digital data to explore the possible influence of usage, acceptance and perceived functioning of the app upon help-seeking behaviours and help-seeking attitudes of participants.

Qualitative analysis will be conducted for the end-of-study qualitative interviews. All interviews will be audio recorded, transcribed verbatim and uploaded to NVivo. The research team will each read through data for emerging themes to develop a coding scheme. When complete, RA will code transcripts to identify major themes. We will use the thematic analysis process to review the transcribed interviews, generate codes, develop themes and finally present the findings in a final report.

ELIGIBILITY:
Inclusion Criteria:

* Aged 17-29 years, inclusive.
* Be enrolled in full-time or part-time studies at one of the participating postsecondary institutions: University of Toronto (St. George and Scarborough campuses), Ryerson University, and George Brown College (all campuses).
* All participants must have functional competency in English.
* Participants must have access to digital devices (smartphone or desktop) compatible with the Thought Spot digital platform.

Exclusion Criteria:

* Individuals who do not have access to a functional mobile device or computer.
* Individuals who are experiencing active suicidality.

Ages: 17 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 481 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The General Help Seeking Questionnaire (change over 6 month trial period) | This scale will be administered at baseline, 3 month and 6 month mark.
  The General Help Seeking Questionnaire is used to measure intentions to seek help from different sources. Future help-seeking intentions are measured by listing a number of potential help sources and asking participants to indicate how likely it is that they would seek help from that source for a specified problem on a seven-point scale ranging from (1) extremely unlikely to seek help to (7) extremely likely to seek help. Higher scores indicate higher intentions for help-seeking. The GHSQ items are scored as a single scale that includes all specific help source options for the specified problem.

SECONDARY OUTCOMES:
Actual Help Seeking Questionnaire (AHSQ) | This scale will be administered at baseline, 3 month and 6 month mark.
  The Actual Help Seeking Questionnaire is used to measure past help seeking. Recent help-seeking behavior is determined by listing a number of potential help sources and asking whether or not help has been sought from each of the sources during a specified period of time for a specified problem. Participants provide a "yes" or "no" response for each help source option that matched those listed in the GHSQ. To provide additional descriptive information and to ensure that participants are responding in the appropriate way, participants are asked to briefly elaborate on the nature of the problem for which help was sought. Participants can also indicate that they have had a problem, but have sought help from no one.
  experiences. A higher total number of instances of help sought from either formal or informal help sources indicates a higher degree of help-seeking behaviour.
Attitudes towards seeking professional psychological help (ATSPPH-SF) | This scale will be administered at baseline, 3 month and 6 month mark.
  The Attitudes Towards Seeking Professional Psychological Help (SF) is used to measure participants process of seeking professional help.This scale measures general attitudes towards seeking professional psychological help for mental health issues. Items are rated on a 4-pointLikert-type scale (3 = Agree,0 = Disagree), where items 2,4,8,9, and 10 are reverse scored. Items are rated from 1 (disagree) to 4 (agree), with five items reversed scored. Scores are summed together with higher scores indicating more positive attitudes toward seeking professional help.
Self-Stigma of Seeking Help Scale (SSOSH) | This scale will be administered at baseline, 3 month and 6 month mark.
  The Self-Stigma of Seeking Help Scale is used to measure change in participants self-stigma of seeking psychological help. Items are rated from 1 (Strongly Disagree) to 5 (Strongly Agree) on a scale of 10 questions. Items 2, 4, 5, 7, and 9 are reverse scored. Because the self- stigma associated with seeking psychological help was hypothesized to keep people from seeking treatment, those who have sought help should have lower SSOSH scores than those who had not. Lower scores (less stigma), therefore, are better outcomes in terms of likelihood to engage in psychological help-seeking. The questions on the SSOSH are scored as a single scale. Items 2, 4, 5, 7, and 9 are reverse scored.
Youth Efficacy/Empowerment Scale - Mental Health (YES-MH) | This scale will be administered at baseline, 3 month and 6 month mark.
  The Youth Efficacy/Empowerment Scale is used to measure change in participants empowerment and efficacy when consuming mental health services. Items are rated from 1 (never or almost never) to 5 (always or almost always), with three items reversed scored. Higher scores from the sum of the subscales represents higher overall youth efficacy/empowerment with respect to mental health. The subscales can be used separately. The sum of their scores yields a score for overall youth efficacy/empowerment with respect to mental health.

CONTACTS AND LOCATIONS:
Overall Officials: David Wiljer, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong HW, Lo B, Shi J, Hollenberg E, Abi-Jaoude A, Johnson A, Chaim G, Cleverley K, Henderson J, Levinson A, Robb J, Voineskos A, Wiljer D. Postsecondary Student Engagement With a Mental Health App and Online Platform (Thought Spot): Qualitative Study of User Experience. JMIR Ment Health. 2021 Apr 2;8(4):e23447. doi: 10.2196/23447. PMID 33797395
- [Derived] Wiljer D, Shi J, Lo B, Sanches M, Hollenberg E, Johnson A, Abi-Jaoude A, Chaim G, Cleverley K, Henderson J, Isaranuwatchai W, Levinson A, Robb J, Wong HW, Voineskos A. Effects of a Mobile and Web App (Thought Spot) on Mental Health Help-Seeking Among College and University Students: Randomized Controlled Trial. J Med Internet Res. 2020 Oct 30;22(10):e20790. doi: 10.2196/20790. PMID 33124984
- [Derived] Kaur A, Isaranuwatchai W, Jaffer A, Ferguson G, Abi-Jaoude A, Johnson A, Hollenberg E, Wiljer D. A Web- and Mobile-Based Map of Mental Health Resources for Postsecondary Students (Thought Spot): Protocol for an Economic Evaluation. JMIR Res Protoc. 2018 Mar 29;7(3):e83. doi: 10.2196/resprot.9478. PMID 29599106
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital — http://www.camh.net/research